CLINICAL TRIAL: NCT01674738
Title: TS Stratified Chemotherapy and VEGF Inhibition in Non-Squamous Non-Small Cell Lung Cancer - Stage IV
Acronym: SELECT-A
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Decision of the Sponsor, as the funding of the study was no longer guaranteed.
Sponsor: Aktion Bronchialkarzinom e.V. (Other)
Collaborators: Roche Pharma AG (Industry); Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ABC-2011-NSCLC-03; 2011-002145-35 (EudraCT Number)
Record Dates: First submitted 2012-08-23; First posted 2012-08-29 (Estimated); Last update posted 2013-10-11 (Estimated); Status verified 2013-10

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: Non Small Cell Lung Cancer; NSCLC Stage IV; Non-Squamous Advanced Non-Small-Cell Lung-Cancer (Stage IV)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Pemetrexed; Cisplatin; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pemetrexed, Cisplatin, Bevacizumab (Experimental): Stratum A
  Interventions: Drug: Pemetrexed; Drug: Cisplatin; Drug: Bevacizumab
- Pemetrexed, Cisplatin, Bevazizumab (Experimental): Stratum B:
  Interventions: Drug: Pemetrexed; Drug: Cisplatin; Drug: Bevacizumab

INTERVENTIONS:
Drug: Pemetrexed — 500 mg/m2 i.v. on day 1 (three-week cycle)
Drug: Cisplatin — 75 mg/m2 i.v. on day 1 (three-week cycle)
Drug: Bevacizumab — 7,5 mg/kg i.v. on day 1 (three-week cycle)

SUMMARY:
This study wants to determine the activity of a first-line treatment related to Thymidylate Synthetase (TS) Expression. Patients with the diagnosis of non-squamous advanced Non-Small-Cell Lung-Cancer (Stage IV) and without evidence of EGFR mutation may be enclosed in this clinical trial.

DETAILED DESCRIPTION:
During the screening procedure tumour specimens obtained by primary biopsy, will be analysed for EGFRmut and immunohistochemically for thymidylate synthetase (TS) expression. Employing the H-Score with a cut-off of 150, EGFR-wt patients will be stratified into a TS low (Stratum A) and TS high (Stratum B) group. This procedure is aiming to provide two equally sized strata.

After stratification according to the TS expression level patients will be treated with a combination of Pemetrexed, Cisplatin and Bevacizumab.

Pemetrexed/Cisplatin/Bevacizumab will be administered for a maximum of 4 cycles. Patients with a complete response (CR), partial response (PR) or stable disease (SD) will continue on maintenance therapy of Pemetrexed and Bevacizumab until disease progression or unacceptable toxicity.

* Duration of treatment/patient: up to 1,5 years
* Follow Up: at least 6 month
* Planned number of patients: 146 treated patients

ELIGIBILITY:
Inclusion Criteria:

* Histological confirmed Non-Small-Cell lung cancer
* Tumor stage IV (UICC 7th Version)
* The following histological tumor types are eligible:

  * Adenocarcinoma (including adenocarcinomas with bronchioloalveolar differentiation)
  * Large Cell carcinoma without neuroendocrine differentiation
  * Mixed Cell Carcinoma without small cell fraction and without predominant squamous cell fraction
  * undifferentiated non-small-cell-carcinoma
* No previous chemotherapy for stage IV NSCLC
* Adjuvant or neoadjuvant chemotherapy for NSCLC must be completed at least one year prior to study enrolment (from end of chemotherapy)
* No previous treatment with Pemetrexed or Bevacizumab
* Patients with prior radiation therapy may be eligible for this study if they meet the following guidelines:

  * Previous radiation therapy is allowed to <25% of the bone marrow (Cristy and Eckerman 1987), but should have been limited and must not have included whole pelvis radiation.
  * Patients must have recovered from the toxic effects of the treatment prior to study enrollment (except for alopecia).
  * Prior thoracic radiotherapy must be completed 30 days before study enrollment.
  * Lesions that have been radiated cannot be included as sites of measurable disease unless clear tumor progression has been documented in these lesions since the end of radiation therapy.
  * Palliative extrathoracic radiotherapy to preexisting lesions may continue on study; however, these lesions may not be included as sites of measurable disease.
* At least 4 weeks since last major surgery
* Age ≥ 18 and ≤ 70 years
* ECOG ≤ 1
* Adequate hematological laboratory parameters:

  * Hemoglobin ≥9 g/dl
  * Neutrophils ≥ 1.500 µl
  * WBC ≥3.000 µl
  * Platelets ≥100.000 µl
* Adequate hepatic laboratory parameters:

  * Total Bilirubin ≤ 1,5 x ULN
  * Alkaline phosphatase ≤ 3 x ULN
  * AST(GOT) < 2,5 ULN in patients without liver metastasis < 5 x ULN in patients with liver metastasis ULN = (upper limit of normal)
  * ALT(GPT) < 2,5 ULN in patients without liver metastasis < 5 x ULN in patients with liver metastasis ULN = (upper limit of normal)
* Adequate renal laboratory parameters:

  * Creatinine Clearance > 50 ml/min
  * Urine dipstick for proteinuria < 2+ Patients discovered to have ≥ 2+ proteinuria on dipstick urinalysis at baseline should undergo a 24-hour urine collection and must demonstrate <1 g of protein in 24 hours
* Normal cardiac function defined by New York Heart Association - NYHA Class I and Class II
* Electrocardiogram without significant signs of cardiac arrhythmias
* Provision of informed consent according to local regulatory requirements prior to any protocol specific treatment.
* Measurable lesion according to RECIST 1.1
* Negative pregnancy test for women of childbearing potential unless they are postmenopausal at baseline. (Postmenopausal women must have been amenorrheic at least for 12 months to be considered of non childbearing potential)
* Women of child bearing potential to be willing to use an acceptable method to avoid pregnancy at least one month before study start. Examples: oral contraceptives (sole application of oral contraceptives is not sufficient), diaphragm pessary, intrauterine device (spiral), condom plus diaphragm pessary plus spermicide.

Exclusion Criteria:

* Histological confirmed predominant squamous cell carcinoma
* Presence of activating EGFR mutations in exons 18-21
* Pregnancy or lactation period
* Have known central nervous system (CNS) disease, other than stable, treated brain metastasis. Stable, treated brain metastasis is defined as metastasis having no evidence of progression or hemorrhage after treatment and no ongoing requirement for dexamethasone, as ascertained by clinical examination and post-treatment brain imaging (CT scan or magnetic resonance imaging [MRI]). Patients should be off corticosteroids for 1 week (7 days) at the time of the post-treatment brain CT/MRI. Anticonvulsants (stable dose) are allowed. Treatment for brain metastases may include whole brain radiotherapy, (stereotactic) radiosurgery (Gamma Knife, linear particle accelerator, or equivalent), or a combination as deemed appropriate by the treating physician, and must have been completed > 8 days prior to Day 1 of Cycle 1. Patients with signs of a fresh bleeding into one or more cerebral metastases or with CNS metastases treated by neurosurgical resection or brain biopsy performed within 8 weeks prior to Day 1 of Cycle 1 will be excluded.
* Evidence of tumor invading or abutting major blood vessels
* Presence of a tracheobronchial fistula
* History of abdominal fistula or fistulisation of urogenital tract, gastrointestinal perforation or intra-abdominal abscess, inflammatory bowel disease, or diverticulitis within 6 months prior to study start
* Other co-existing malignancies or malignancies diagnosed within the last 5 years with the exception of a CIS of the cervix, non-melanomatous skin cancer, stable chronic lymphatic leukaemia, non-muscle invasive bladder cancer or surgically treated or irradiated prostate cancer with no signs of recurrence for one year. Patients with other malignancies curatively treated and free of disease for at least 5 years will be discussed with the Principal Investigator (LKP) before inclusion.
* Treatment with an investigational new drug, currently or within the last 28 days, and/or participation in another clinical trial, currently or during the last 12 weeks, and/or previous participation in this study.
* History or presence of a mental disease or condition such as to interfere with the patient's ability to understand the requirements of the study and the intake of study medication according to study protocol.
* Patients with any clinically significant disease that in the opinion of the investigator is likely to put the patient at risk or to interfere with the evaluation of the patient's safety and of the study outcome. This includes, but is not limited to:

  * Immediate need for therapeutic intervention (e.g.: upper inflow congestion or poststenotic pneumonia).
  * Clinically significant cardiac disease (e.g. right-sided heart failure, symptomatic coronary artery disease and cardiac arrhythmias not well controlled with medication) or myocardial infarction within the last 6 months.
* Have a history of hypertension, unless hypertension is well controlled upon study entry (<150/90 mm Hg) and the patient is on a stable regimen of antihypertensive therapy. Patients should not have any prior history of hypertensive crisis or hypertensive encephalopathy.
* Non healing wound, ulcer or bone fracture
* Fresh thrombosis (within the last two weeks) under full dose therapy with anticoagulants.
* History of thrombotic disorders within the last 6 months prior to entry.
* Current or recent (within 10 days of first dose of study medication) full-dose oral or parenteral anticoagulants, or thrombolytic agents for therapeutic purposes.
* Prophylactic use of anticoagulants is allowed; international normalized ratio (INR) should be <1.5 at study enrollment.
* Current or recent (within 10 days of first dose of study medication) use of ASS - Dosage > 325 mg/day
* Current or recent (within 10 days of first dose of study medication) use of Plavix/Clopidogrel, at doses >75 mg/d, dipyramidole, ticlopidine, cilostazol,
* Hemorrhagic diathesis, Hemophilia A, Hemophilia B
* Implantation of a central vein catheter (Implanted port catheter) within 24 h prior to application of study medication
* Have a history of gross hemoptysis (bright red blood of ½ teaspoon per episode of coughing) <3 months prior to enrollment or history or evidence of inherited bleeding diathesis or coagulopathy with the risk of bleeding.
* Peritoneal carcinomatosis.
* Pleural effusion with the need of therapeutic pleurodesis
* Ascites with the need of intervention
* Any other uncontrolled infection
* Organ allograft
* Hardness of hearing that interferes with daily life
* Sensory Neuropathy > grade I (CTCAE Version 4.0 )
* Alcohol and drug abuse
* Known hypersensitivity to any of the study drugs
* Have a history of a serious reaction to a monoclonal antibody. Patients with known hypersensitivity to Chinese hamster ovary cell products or other recombinant human antibodies are not eligible.
* Have received a recent (within 30 days of enrollment) or are receiving concurrent yellow fever vaccination
* Have had major surgery, open biopsy, or significant traumatic injury within 28 days prior to study enrollment, or anticipate the need for major surgical procedure during the course of the study.
* Patients with creatinine clearance 45-79 ml/min must be able to interrupt NSAIDs 2 days before (5 days for long-acting NSAIDs ), the day of, and 2 days following administration of pemetrexed.
* Are unable or unwilling to take folic acid, vitamin B12 supplementation, or corticosteroids.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
Progression free survival | Recruitment period 1,5 years, observation period 2 years

SECONDARY OUTCOMES:
Overall survival | Recruitment period 1,5 years, observation period 2 years
Quality of life | Screening, day 1, end of cycle 1, end of treatment (for each patient)
Response rate | Screening, prior to cycle 3, end of cycle 4, evry 6 weeks after end of cycle 4, end of treatment (for each patient)
Molecular investigations | Day 1, prior to cycle 3, end of cycle 4, end of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Gunther Wiest, MD, Principal Investigator — Asklepios Klinik Harburg, D-21075 Hamburg, Germany; Prof. Dr. Martin Wolf, MD, Study Chair — Klinikum Kassel GmbH, D-34125 Kassel; Dr. Monika Serke, MD, Study Chair — Lungenklinik Hemer, D-58675 Hemer, Germany; Prof. Dr. Michael Thomas, MD, Study Chair — Thoraxklinik Heidelberg, D-69126 Heidelberg, Germany; Rudolf M. Huber, MD, Study Chair — Klinikum der Universität München, D-80336 München, Germany